CLINICAL TRIAL: NCT03588858
Title: Child Labour at Al-Sadat Neighborhood, Assiut City
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hisham Ragab Ali (Other)
Responsible Party: Sponsor-Investigator, Hisham Ragab Ali, Physician at Public Health and Community Medicine department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Child labour at Assiut city
Record Dates: First submitted 2018-04-11; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Work-Related Condition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: structured interview questionnaires — * Module (1): Socio-demographic characteristics
  * Module (2) :Occupational history
  * Module (3): Presence of work related injuries and diseases by history and observation.
  * Module (4): Food frequency questionnaires (FFQ) during the past week.
  * Module (5): Mental health screening: Self-reporting questionnaire 20 questions for assessment of mental health status of children.

SUMMARY:
General objective: To promote proper health status of working children in Assiut city.

Specific objectives:

1. To describe the socio-demographic characteristics of children working in car repair workshops in Al-Sadat area of Assiut city.
2. To describe the work environment.
3. To identify work related injuries and diseases among those working children.

DETAILED DESCRIPTION:
Study population: Children working in car repair workshops in Al-Sadat area of Assiut city. Male children aged from 5 to 17 years will be included in this study.

Instrument: Data collection will be performed by using structured interview questionnaires. The questionnaire used for data collection will cover the following modules:

* Module (1): Socio-demographic characteristics (for example: age, family size, family residence, education and occupation of the parents, number of sibling, family income, etc).
* Module (2) :Occupational history : (Housing conditions and occupational features; age at the beginning of working, duration of working, working hours/day, weekend vacation, weekly income, causes of child work, nature of work, work hazards, type of exposure, health habits and practices such as smoking in addition to causes of school dropout…. etc)
* Module (3): Presence of work related injuries and diseases by history and observation.
* Module (4): Food frequency questionnaires (FFQ) during the past week: It will show the diet of working children if have a healthy and nutritious pattern or not.
* Module (5): Mental health screening: Self-reporting questionnaire 20 questions for assessment of mental health status of children.
* After collection of data the children will subjected to the following investigations:

HB level measurements - anthropometric measurements (weight and height) - pulmonary function tests (spirometry) and hearing level assessment by audiometry will be done only for children more than 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Children working in car repair workshops in Al-Sadat area of Assiut city. Male children aged from 5 to 17 years

Exclusion Criteria:

* Children outside the age range (below 5 years),
* Female children

Ages: 5 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male children aged from 5 to 17 years will be included in this study.
Study Population: The study will be conducted at the workshops of car repair in Al-Sadat area of Assiut city. The number of these workshops is 130 and the number of working children in these workshops about 150 child.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level measurements by using Mission Hb Hemoglobin Meter | Baseline
  gm/dl

SECONDARY OUTCOMES:
measurements (weight by weighing scale and height by height scale) | Baseline
  weight in kilograms and height in centimeters will be combined to report Body Mass Index in kg/m^2).

OTHER OUTCOMES:
pulmonary function tests | Baseline
  by using spirometry device

CONTACTS AND LOCATIONS:
Overall Officials: Sabra Ahmed, MD, Principal Investigator — Assistant professor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ILO. What is child labour, International Labour Organization